CLINICAL TRIAL: NCT00034424
Title: Multidisciplinary Etiologic Study of Familial Testicular Cancer
Brief Title: Cause of Familial Testicular Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020178; 02-C-0178; NCT00039598 (obsolete NCT alias)
Record Dates: First submitted 2002-04-27; First posted 2002-04-29 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-05-23

CONDITIONS: Testicular Cancer
Keywords: Genetics; Hereditary; Screening; Behavioral; Familial Testicular Germ Cell Tumor; Natural History; Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms; Behavior

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: individuals from families with familial TGCT

SUMMARY:
Background:

People with a family history of testicular cancer may be at increased risk for the disease.

Genetic and clinical studies of patients with testicular cancer and their family members may help clarify the cause of the disease and identify clinical features.

Objectives:

To characterize the clinical features of testicular cancer.

To identify genes that may lead to increased risk of the disease.

To examine emotional and behavioral issues of members of families at increased risk of the disease.

Eligibility:

Males and females from a family with at least two cases of testicular cancer in blood relatives.

Males with testicular cancer in both testicles.

Males with testicular cancer who have an identical twin.

Participants must be at least 12 years of age.

Design:

Participants may take part in Part 1 or Parts 1 and 2 of this 2-part study.

Part 1 participants:

* Provide a blood or cheek cell sample to obtain DNA for gene studies.
* Provide permission for researchers to obtain their medical records for review.
* Complete questionnaires about their personal and family medical history, exposure to factors that might influence the risk of testicular cancer, and their feelings about being a member of a family in which several members have testicular cancer.
* These data are collected from participants in their home communities.

Part 2 participants:

* All participants provide a medical history, have a complete physical examination, including routine lab tests, and have an ultrasound test of the abdomen to look at the kidneys.
* Males have an ultrasound test of the testicles and scrotum.
* Females have an ultrasound test of the pelvis to look at the ovaries, uterus and fallopian tubes.
* Males 18 years of age and older provide a semen sample.
* Some participants have computed tomography (CT) scanning of the chest, abdomen and pelvis instead of kidney ultrasound. Children under 18 years of age may have magnetic resonance imaging (MRI) instead of CT.
* These data are collected from participants during a 2-day visit to the NIH Clinical Center in Bethesda, MD. Travel costs are covered by the protocol.

DETAILED DESCRIPTION:
BACKGROUND:

Testicular germ cell tumor (TGCT) is the most common cancer in men aged 20-35, with an increasing incidence since the mid-twentieth century.

A family history of TGCT is associated with an increased risk of the disease.

Evidence suggests that there is genetic heterogeneity in familial TGCT, thereby creating opportunities for both new susceptibility gene discovery and searching for genotype/phenotype/cancer correlations.

Search for genitourinary developmental anomalies and for testicular intraepithelial neoplasia (TIN) cells which are thought to be the precursor of the vast majority of TGCT could help clarify the etiology and identify clinical features.

This project is both etiologic and clinical in its focus, and its goal is to acquire a comprehensive understanding of both the genetic and non-genetic factors which contribute to the risk of familial TGCT.

OBJECTIVES:

Ascertain new families with familial testicular germ cell tumors.

Characterize the clinical features of familial TGCT.

Determine the underlying genetic mechanism for susceptibility to TGCT in families; one specific goal is to confirm, and then to clone, the hereditary testicular cancer gene which has been mapped to chromosome Xq27.

Evaluate various parameters related to psychosocial and behavioral issues resulting from being a member of a family at increased risk of TGCT.

ELIGIBILITY:

A single family member with bilateral testicular cancer.

Individuals of both genders from a family with at least two cases of documented GCT in blood relatives (at least one of which is testicular in origin) and with at least one of the GCT cases in their family willing to participate in the study.

Men with a history of TGCT who have a monozygotic twin brother (the unaffected identical sibling must also agree to participate).

Families will be deemed ineligible if critical informative family members lacking surviving spouses and children are unable to provide germ line DNA

Minor children under age 12 will not be eligible for study participation.

DESIGN:

International collaboration between NCI's Clinical Genetics Branch and the International Testicular Cancer Linkage Consortium (ITCLC), via contribution of DNA.

Non-randomized cohort study with an estimated accrual of 75 and 100 new TGCT families over a period of 5 years and approximately 40 families willing to visit the NIH Clinical Center.

Individuals and family members will be asked to contribute baseline questionnaires as well as questionnaires regarding lifestyle, feelings, attitudes and behavior that relate to being part of a high-risk family, and DNA for gene mapping and cloning efforts.

Detailed, in-person, etiologically-oriented evaluation at the NIH Clinical Center includes a comprehensive history and physical examination, laboratory testing, and ultrasound imaging of the kidneys and gonads to identify the clinical features and seek clinically occult TGCT and TIN. CT imaging studies of the chest, abdomen, and pelvis will be performed when indicated.

Study participants will be monitored prospectively for the development of outcomes of interest by means of periodic mail and/or telephone contact. Cancer outcomes will be documented through review of medical, vital, and pathology records. Tumor tissue will be obtained whenever feasible.

As of December 2021, research activities under this protocol are limited to the follow-up collection of medical records and questionnaires from consented individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:

Study population:

Patients must be members of families with familial TGCT as defined below.

Definition of familial TGCT:

The criterion establishing familial TGCT is the presence of:

-at least two cases of documented GCT in blood relatives (at least one of which is testicular in origin),

OR

* a single family member with bilateral testicular cancer,
* men with a history of TGCT who are one in a set of identical siblings will also be included in the study.

Case definition:

A case will be determined to have TGCT according to the following criteria:

* Pathologic confirmation of a germ cell derived tumor arising in the testis. Extragonadal germ cell tumors will also be included.
* Germ cell derived histologies including: seminoma, germinoma, embryonal carcinoma, endodermal sinus (yolk sac) tumor, gonadoblastoma, choriocarcinoma, teratoma, and mixed germ cell tumor.
* A case will be determined to have TIN on the basis of pathologic confirmation of intratubular malignant germ cells (ITMGCs) as defined by Burke and Mostofi.

Individuals from participating families who are eligible for this study include:

i) all TGCT cases;

ii) all GCT cases (including those of ovarian or extra-gonadal sites);

iii) all first-degree relatives of each GCT case;

iv) the spouse(s) of every case if the spouse and case had children who are participating in the study;

v) any blood relative not included in (ii - iii) above who genetically links two cases; and

vi) any blood relative with cancer other than GCT

vii) family members as described in i) - v) above must be age 12 or greater in order to participate

EXCLUSION CRITERIA:

Families will be deemed ineligible for participation in this study if:

There are not at least two confirmed cases of GCT in the family, (at least one of which is testicular in origin), unless there is a family member with bilateral testicular cancer;

Deceased TGCT cases lacking both archival sources of tissue for DNA extraction AND lacking surviving spouses and children who are willing to participate in the study (the unavailability of such persons prohibits inferring the genotype of the deceased individual with TGCT);

Critical informative family members are unwilling to participate (i.e., unwilling to provide written informed consent);

Ages: 12 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A non-randomized cohort study of individuals from families with a significant history of testicular cancer.
Sampling Method: Non-Probability Sample
Enrollment: 749 (Actual)
Dates: Start 2003-01-13 (Actual)

PRIMARY OUTCOMES:
Families with Familial Testicular Germ Cell Tumors | Ongoing
  Ascertain new familiies with FTGCTs
Clinical Features | Ongoing
  Characterize the clinical features of familial TGC
Genetic Mechanisms | Ongoing
  Determine the underlying genetic mechanism for susceptibility to TGCT in families
Psychosocial Factors | Ongoing
  Evaluate psychosocial issues related to FGCT

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Stewart, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Azevedo MF, Horvath A, Bornstein ER, Almeida MQ, Xekouki P, Faucz FR, Gourgari E, Nadella K, Remmers EF, Quezado M, de Alexandre RB, Kratz CP, Nesterova M, Greene MH, Stratakis CA. Cyclic AMP and c-KIT signaling in familial testicular germ cell tumor predisposition. J Clin Endocrinol Metab. 2013 Aug;98(8):E1393-400. doi: 10.1210/jc.2012-2838. Epub 2013 Jun 14. PMID 23771924
- [Background] Chung CC, Kanetsky PA, Wang Z, Hildebrandt MA, Koster R, Skotheim RI, Kratz CP, Turnbull C, Cortessis VK, Bakken AC, Bishop DT, Cook MB, Erickson RL, Fossa SD, Jacobs KB, Korde LA, Kraggerud SM, Lothe RA, Loud JT, Rahman N, Skinner EC, Thomas DC, Wu X, Yeager M, Schumacher FR, Greene MH, Schwartz SM, McGlynn KA, Chanock SJ, Nathanson KL. Meta-analysis identifies four new loci associated with testicular germ cell tumor. Nat Genet. 2013 Jun;45(6):680-5. doi: 10.1038/ng.2634. Epub 2013 May 12. PMID 23666239
- [Background] Schumacher FR, Wang Z, Skotheim RI, Koster R, Chung CC, Hildebrandt MA, Kratz CP, Bakken AC, Bishop DT, Cook MB, Erickson RL, Fossa SD, Greene MH, Jacobs KB, Kanetsky PA, Kolonel LN, Loud JT, Korde LA, Le Marchand L, Lewinger JP, Lothe RA, Pike MC, Rahman N, Rubertone MV, Schwartz SM, Siegmund KD, Skinner EC, Turnbull C, Van Den Berg DJ, Wu X, Yeager M, Nathanson KL, Chanock SJ, Cortessis VK, McGlynn KA. Testicular germ cell tumor susceptibility associated with the UCK2 locus on chromosome 1q23. Hum Mol Genet. 2013 Jul 1;22(13):2748-53. doi: 10.1093/hmg/ddt109. Epub 2013 Mar 5. PMID 23462292
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0178.html